CLINICAL TRIAL: NCT03365843
Title: Montage- Enhanced Sternal Closure to Accelerate Post-Operative Recovery
Brief Title: Montage-Enhanced Sternal Closure
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Calgary (Other)
Collaborators: Abyrx, Inc. (Industry)
Responsible Party: Principal Investigator, Dr. Paul Fedak, Professor and Cardiac Surgeon, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: REB17-1399
Record Dates: First submitted 2017-10-26; First posted 2017-12-07 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Sternal Closure
Keywords: Cardiac surgery; Sternal closure

STUDY DESIGN:
Intervention Model Description: Randomized, single centre, double-blind clinical study
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The participants, study coordinator and care-givers are blinded to the assigned treatment arm. Participants may be able to guess which treatment group they have been assigned. This will be assessed at the end of the study by asking participants to identify the group to which they think they have been assigned.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Montage bone putty (Experimental): Sternal closure with conventional wire cerclage plus Montage bone putty
  Interventions: Device: Montage bone putty; Other: Conventional Sternal Closure
- Conventional Sternal Closure (Active Comparator): Conventional wire cerclage sternal closure only -- standard care.
  Interventions: Other: Conventional Sternal Closure

INTERVENTIONS:
Device: Montage bone putty — Application of bone putty on cut sternal surfaces prior to application of conventional wires for closure of sternum during cardiac surgery.
  Arms: Montage bone putty
Other: Conventional Sternal Closure — Closure of sternum with standard wire cerclage.

SUMMARY:
Post-operative recovery after cardiac surgery is influenced by early sternal bone stability. Traditional sternal closure of median sternotomy usually entails the use of 6-10 stainless steel wires. Augmenting sternal closure with techniques to enhance early bone stability should accelerate functional recovery from cardiac surgery thereby reducing post-operative pain, decreasing the need for narcotics, improving breathing and chest wall mechanics, stimulating early mobility and expediting hospital discharge.

This study is a randomized, single-centre, double-blind clinical study comparing the effects of Montage bone putty plus conventional wire closure vs conventional wire closure only on the post-operative recovery of cardiac surgery patients with full medial sternotomy.

DETAILED DESCRIPTION:
Patients undergoing cardiac surgery who are participating in the study will be randomized to either conventional wire cerclage or conventional wire closure plus the use of Montage bone putty. Patients will be followed post-operatively Day 3, 5 and at discharge as well as weeks 2, 4, 6 and months 3, 6 and 12.

Each visit will include: Pain assessment, wound assessment, sternal assessment, analgesic/antibiotic use, spirometry testing, quality of life questionaries (EQ-5D/HAQ) and determination of any adverse events. Chest x-rays will done at discharge and 3, 6, and 12 months to look at sternal healing.

This pilot study will include a total of 65 patient (40 conventional + putty / 20 conventional/ 5 initial open label with putty).

ELIGIBILITY:
Inclusion Criteria:

* undergoing non-emergent cardiac surgery ( cabg only or one valve procedure)
* full median sternotomy approach, with or without cardiopulmonary bypass
* English speaking
* geographically accessible
* written consent

Exclusion Criteria:

* Recent CPR
* previous cardiac surgery
* emergency surgery ( within 24 hrs of assessment)
* chronic lung disease
* history of bleeding disorder
* currently taking Vitamin E supplements
* recent antiplatelet therapy
* excessively poor baseline health-related quality of life or physical functioning
* previous radiotherapy to chest, or on immunosuppressive drugs or current immunosuppressive condition
* active significant systemic infection, history of recurrent infections,
* cognitive impairment ( confusion, dementia, Alzheimer's, current substance abuse)
* history of malignancy within the past year
* recent history of significant alcohol or drug abuse
* females who are pregnant, nursing, or child bearing potential who are not practicing a highly reliable birth control method
* postsurgical life expectancy of less than 90 days
* moderate to severe pectus deformity
* participation in another study

Ages: 19 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Recovery of Respiratory Function | Intervention to 6 weeks post-operative
  The recovery of pulmonary functional capacity as measured by the return of forced vital capacity (FVC) to 80% or greater of the pre-operative baseline FVC measurement.
Radiographic Sternal Integrity | Intervention to 12 months post-operative
  No radiographic evidence of bony instability as assessed through serial chest x-rays
Sternal Revision | Intervention to 12 months post-operative
  Absence of device (wire or Montage bone putty) removal, revision or reoperation occurring over first 12 months post-operative.

SECONDARY OUTCOMES:
Post-operative Pain Assessment | Baseline to 12 months post - operative.
  Severity of post-operative pain (survey score and analgesic use) comparing treatment vs control groups
Rate of post-operative recovery | Baseline to 12 months post-operative
  Rate of post-operative recovery as measured by health related quality of life (EQ5D) standardized assessment tool
Rate of post-operative recovery | Baseline to 12 months post-operative
  Rate of post-operative recovery as measured by physical functioning (HAQ) standardized assessment tool
Sternal Wound Infections | Baseline to 12 months post-operative
  Frequency of sternal wound infections (superficial and deep) between groups
Pulmonary Complications | Baseline to 6 weeks post-operative
  Post-operative pulmonary complications between groups
Health Services resource usage | Baseline to 12 months post-operative
  To compare the burden of health services resource usage between groups (total cost estimate)

CONTACTS AND LOCATIONS:
Overall Officials: Paul WM Fedak, MD, PhD, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vasanthan V, Fatehi Hassanabad A, Kang S, Dundas J, Ramadan D, Holloway D, Adams C, Ahsan M, Fedak PWM. Novel hardening bone putty enhances sternal closure and accelerates postoperative recovery. J Thorac Cardiovasc Surg. 2023 Nov;166(5):e430-e443. doi: 10.1016/j.jtcvs.2022.09.016. Epub 2022 Sep 17. PMID 36272766